CLINICAL TRIAL: NCT00982345
Title: Brain Imaging of Quetiapine Response in Anxious Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0901-13
Record Dates: First submitted 2009-09-21; First posted 2009-09-23 (Estimated); Results first posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Major Depression
Keywords: Depression; Anxiety; Seroquel; Quetiapine; fMRI; pictures
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Anxiety Disorders | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label Quetiapine (Other): Open-label Quetiapine XL 50 - 400 mg daily treatment 8 weeks
  Interventions: Drug: quetiapine (Seroquel XR)

INTERVENTIONS:
Drug: quetiapine (Seroquel XR) — Seroquel XR (starting dose 100mg and increased up to 400 mg as tolerated) treatment.
  Other Names: Seroquel XR

SUMMARY:
The purpose of this study is to find out what parts of the brain have increased or decreased connectivity when people are depressed and how Seroquel extended release (XR) changes this connectivity in depressed patients. The genetic samples collected are to look at variation in a gene (serotonin transporter gene), which affects the functioning of the chemical serotonin in the brain.

DETAILED DESCRIPTION:
This study will measure the activity and connectivity in different parts of the brain, while the patients are seeing some pictures, using Magnetic Resonance Imaging (MRI) scan. For this study three MRI scans will be conducted. One before the patient begins on any medication, one during the study after 3 weeks of treatment and one after six more weeks of treatment with seroquel.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* A diagnosis of Major Depressive Episode by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV)
* Females or Males aged 18 - 60 years
* Female subjects of childbearing potential must be using a reliable method of contraception and have a negative serum human chorionic gonadotropin (HCG) test at enrollment
* Able to understand and comply with the requirements of the study
* 17-item Hamilton Depression Rating Scale (HDRS) score > 15
* Hamilton Anxiety Scale (HAM-A) score > 15
* Satisfy criteria to undergo an MRI scan based on MRI screening questionnaire
* Able to be managed as outpatients for initial assessment and during treatment as ascertained by the following:

  * Symptoms not worsening by more than 10 points on the HDRS during the course of the study.
  * No danger to self or others.

Exclusion Criteria:

* Pregnancy or lactation
* Meeting DSM-IV criteria for schizophrenia, schizophreniform disorder, schizoaffective disorder, atypical psychosis, mental retardation, or organic mental (including organic mood) disorder
* Subjects who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Known intolerance or lack of response to quetiapine fumarate, as judged by the investigator
* Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
* Use of any of the following cytochrome P450 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
* Substance or alcohol dependence at enrollment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
* Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within four weeks prior to enrollment
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical illness (angina pectoris, hypertension) as judged by the investigator
* Involvement in the planning and conduct of the study
* Previous enrollment or randomization of treatment in the present study.
* Participation in another drug trial within four weeks prior enrollment into this study or longer in accordance with local requirements
* A subject with Diabetes Mellitus; people who develop hyperglycemia will be removed from the study
* An absolute neutrophil count (ANC) of 1.5 x 109 per liter
* Use of psychotropics in the past two weeks. If on fluoxetine in the past, then should not have been on this medication for four weeks.
* History of lack of response to Quetiapine extended release.
* Acutely suicidal or homicidal or requiring inpatient treatment.
* Metallic implants.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Anand, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Adult Psychiatry Clinic, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Seroquel XR: Seroquel XR (quetiapine) starting dose 50 mg and increased up to 400 mg as tolerated) treatment.
Period: Overall Study
Arm/Group | Seroquel XR
Started | 20
Completed | 18
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Quetiapine: quetiapine (Seroquel XR) : Seroquel XR (starting dose 100mg and increased up to 400 mg as tolerated) treatment.
Arm/Group | Quetiapine
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: 17-item Hamilton Depression Rating Scale (HDRS)
Description: Standard 17-item rating scale for depression used in clinical trials. A score of 0-7 is considered to be normal. 8 - 13 mild depression. Scores of 20 or higher indicate moderate, severe, or very severe depression, and are usually required for entry into a clinical trial. Range of score: 0 - 50.
Time Frame: Started: March 2009 Ending March 2011
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine
Number analyzed (Participants) | 20
units on a scale
  Baseline 17-item HDRS | 20 (3)
  Post-treatment at 8 weeks 17-item HDRS | 8 (6)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 12 weeks.
Arm/Group | Quetiapine
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 18/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine (N=20)
fatigue (Nervous system disorders) | 16
Irritability (Nervous system disorders) | 3
dizziness (Nervous system disorders) | 7
increased sleep (Nervous system disorders) | 15
headache (Nervous system disorders) | 4
dry mouth (Nervous system disorders) | 12
urinary frequency (Renal and urinary disorders) | 2
blurred vision (Nervous system disorders) | 1
indigestion (Gastrointestinal disorders) | 2
constipation (Gastrointestinal disorders) | 6
increased appetite (Gastrointestinal disorders) | 5
decreased sleep (Nervous system disorders) | 2
abdominal pain (Gastrointestinal disorders) | 4
fluid retention (Vascular disorders) | 1
twitching (Nervous system disorders) | 3
sweating (Nervous system disorders) | 2
hand dryness (Skin and subcutaneous tissue disorders) | 1
nausea (Gastrointestinal disorders) | 3
tremor (Nervous system disorders) | 1
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1
increased thirst (Gastrointestinal disorders) | 1
hives (Skin and subcutaneous tissue disorders) | 1
nose congestion (Respiratory, thoracic and mediastinal disorders) | 1
fainting (Nervous system disorders) | 1
decreased appetite (Gastrointestinal disorders) | 2
DIARRHEA (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
Open label study. Small sample

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No